CLINICAL TRIAL: NCT07307963
Title: Sensitivity of the Load-Velocity Relationship Variables to Discriminate the Level of Fatigue Induced by Multiple Sets of the Smith-Machine Squat Exercise
Brief Title: Sensitivity of Load-Velocity Measures for Detecting Fatigue During Smith-Machine Squats
Acronym: SLV
Status: Completed | Type: Observational
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Deniz ŞENTÜRK, Assistant Professor, PhD, Istanbul Gelisim University
Other Study IDs: 2024/04/67
Record Dates: First submitted 2025-11-27; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Neuromuscular Fatigue; Load-velocity Variables
Keywords: resistance training; fatigue; velocity-based training
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Condition: Control Protocol Arm:
  Participants completed no exercise between the pre- and post-session load-velocity tests.
  Interventions: Other: Control Protocol (No Training)
- Moderate-Fatigue Protocol: Participants performed 5 sets of the Smith-machine squat at 70% of their 1RM, completing half of the maximum possible number of repetitions in each set. This protocol was designed to induce a moderate level of fatigue while avoiding complete muscular failure.
  Interventions: Other: Moderate-fatigue
- High-Fatigue Protocol: In the high-fatigue protocol, participants performed five sets of Smith-machine squats at 70% of their 1RM, completing each set to muscular failure. In every set, participants continued lifting until they could no longer complete a full repetition with proper technique. This protocol was designed to induce a high level of neuromuscular fatigue and to test the sensitivity of load-velocity variables under maximal fatigue conditions.
  Interventions: Other: High-fatigue

INTERVENTIONS:
Other: Control Protocol (No Training) — This intervention consists of no training or exercise during the session. Participants assigned to the control arm rest for the entire duration between the pre-session and post-session load-velocity assessments. No fatigue-inducing activity, resistance exercise, or additional intervention is administered, allowing all observed changes to reflect normal variation without training-related fatigue.
  Groups: Control Condition
Other: Moderate-fatigue — Participants performed five sets of Smith-machine squats at 70% of their 1-repetition maximum (1RM), completing half of the maximum possible repetitions in each set. This protocol was designed to induce a moderate level of neuromuscular fatigue without reaching complete exhaustion.
  Groups: Moderate-Fatigue Protocol
Other: High-fatigue — This intervention involves no training or fatigue-inducing activity. Participants do not perform any squat sets between the pre- and post-session incremental loading tests. This condition serves as a baseline to determine natural variations in load-velocity measures, thereby eliminating the influence of exercise-induced fatigue.
  Groups: High-Fatigue Protocol

SUMMARY:
The purpose of this study is to determine whether load-velocity (L-V) relationship variables (L0, v0, and Aline) are sensitive indicators of fatigue produced by different squat fatigue protocols. The study aims to answer how accurately these L-V measures reflect changes in performance, particularly changes in one-repetition maximum (1RM), after varying levels of induced fatigue. Twenty-eight resistance-trained men completed three sessions involving different fatigue protocols or no training. L-V variables measured before and after each protocol were compared. The findings will help determine whether L-V relationship parameters can be used as practical and sensitive tools for monitoring fatigue during resistance training.

DETAILED DESCRIPTION:
This study investigates how different levels of fatigue influence the parameters of the load-velocity (L-V) relationship during the Smith-machine squat exercise. After an initial familiarization and baseline testing session used to establish 1-repetition maximum (1RM) and to perform a repetition-to-failure test at 70% 1RM, participants completed three separate experimental sessions. Each session implemented a distinct fatigue protocol, and all protocols were performed between two incremental loading tests to determine pre-session and post-session L-V profiles.

The moderate-fatigue condition consisted of five sets at 70% 1RM, with participants performing half of their maximal possible repetitions per set. The high-fatigue condition required five sets performed to volitional failure using the same relative load. A control condition with no exercise was also included to establish non-fatigue reference values. L-V variables of interest included L0, v0, and Aline (calculated as L0 × v0 / 2). These variables were compared across conditions to determine their responsiveness to increasing levels of fatigue and their association with changes in neuromuscular performance, particularly reductions in 1RM strength.

ELIGIBILITY:
Inclusion Criteria:

Healthy males aged 18-40 years.

Resistance-trained (minimum 2 years of regular lower-body resistance training and ≥2 sessions/week).

Able to perform a proper smith-machine back squat with correct technique.

1-RM smith-machine squat measurable and ≥ bodyweight (or specify threshold used in study).

No musculoskeletal injury of lower limbs or back in the past 6 months.

Not using performance-enhancing drugs or anabolic steroids for the past 12 months.

Willing and able to attend all testing and training sessions and provide written informed consent.

Exclusion Criteria:

Any cardiovascular, pulmonary, metabolic, or neurological disease contraindicating intense exercise.

Recent (≤6 months) lower-extremity or spinal surgery or acute injury.

Current musculoskeletal pain or injury that limits squat performance.

Use of medications that affect neuromuscular performance (e.g., systemic corticosteroids) or stimulant drugs.

Regular participation in structured lower-body rehabilitation programs.

Failure to complete familiarization or preliminary 1-RM testing.

Inability or unwillingness to provide informed consent or follow study procedures.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty-eight physically trained males, with an average age of 23.3 years (standard deviation [SD]: 3.0 years; range: 20-36 years), willingly enrolled in this research endeavor. The participants exhibited a mean body mass of 78.1 kg (SD: 9.3 kg), a body height of 177.2 cm (SD: 3.3 cm), and a one-repetition maximum (1RM) for smith-machine squat (SMS) exercise of 150.9 kg (SD: 12.5 kg). All subjects possessed prior RT experience, averaging 5.0 years (SD: 2.6 years), and demonstrated proficiency in executing the SMS exercise during the familiarization session.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Change in Theoretical Maximal Load (L0) Derived From the Load-Velocity Relationship | Baseline (pre-session) and immediately post-session (within 15 minutes)
  Difference in theoretical maximal load (L0, kg) derived from the load-velocity relationship between baseline (pre-session) and immediately post-session incremental loading tests.

SECONDARY OUTCOMES:
Change in Theoretical Maximal Velocity (v0) Derived From the Load-Velocity Relationship | Baseline (pre-session) and 15 minutes post-session
  Difference in theoretical maximal velocity (v0, m/s) derived from the load-velocity relationship between baseline (pre-session) and immediately post-session incremental loading tests.
Change in Area Under the Load-Velocity Relationship Line (Aline) | Baseline (pre-session) and immediately post-session (within 15 minutes)
  Difference in area under the load-velocity relationship line (Aline, calculated as L0 × v0 / 2) between baseline (pre-session) and immediately post-session incremental loading tests.
Change in One-Repetition Maximum (1RM) in the Smith-Machine Squat | Baseline (pre-session) and immediately post-session (within 15 minutes)
  Difference in one-repetition maximum (1RM, kg) in the smith-machine squat between baseline (pre-session) and immediately post-session incremental loading tests.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Şentürk, PhD, Principal Investigator — Istanbul Gelisim University
Locations (1):
- İstanbul Gelişim Üniversity, Istanbul, avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared after de-identification. Data will be available to qualified researchers upon reasonable request for academic purposes. Access will be provided following publication of the primary results. Researchers will be required to submit a brief proposal describing the intended use of the data, and data will be shared through secure, controlled access. No identifiable information will be released.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data and supporting documents will become available 6 months after publication of the study results and will remain available for 5 years.
Access Criteria: Individual participant data (IPD) will be shared in anonymized form with qualified researchers for scientific purposes. The shared data will include de-identified performance measurements, load-velocity variables, and outcome measures relevant to the study.
URL: https://zenodo.org/records/17572347